CLINICAL TRIAL: NCT04886453
Title: Evaluation of Non-opioid Balanced General Anesthesia in Cardiac Surgery With Extracorporeal Circulation: a Randomized, Controlled, Multicenter Superiority Trial
Acronym: OFACAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOUHEMAD PHRCI 2019
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Opioid-free Anesthesia; Cardiac Surgery
MeSH Terms: interventions — Morphine; Data Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: Balanced general anesthesia without morphine; Other: Data collection; Other: Assessment of pain; Other: Recovery quality score
- Controle (Active Comparator)
  Interventions: Drug: Standard general anesthesia balanced with morphine; Other: Data collection; Other: Assessment of pain; Other: Recovery quality score

INTERVENTIONS:
Drug: Balanced general anesthesia without morphine — Balanced general anesthesia without morphine
  Arms: Intervention
Drug: Standard general anesthesia balanced with morphine — Standard general anesthesia balanced with morphine
  Arms: Controle
Other: Data collection — Data collection
Other: Assessment of pain — visual analog scale
Other: Recovery quality score — QoR15 questionnaire

SUMMARY:
Opioid-free anesthesia (OFA) is a general anesthesia based on the use of hypnotics and non-opioid analgesics (lidocaine, ketamine, dexamethasone, esmolol). This technique has been used for the past 10 years, during which randomized and non-randomized studies have demonstrated a number of positive effects on cardiac function:

* better analgesia and decreased postoperative morphine consumption,
* better respiratory function,
* better hemodynamic stability,
* better postoperative cognitive function.

The hypothesis of the present study is that the use of OFA during cardiac surgery is associated with:

* Improved intraoperative hemodynamic stability
* A decrease in the incidence of postoperative complications
* A reduction in intensive care and hospital length of stay

ELIGIBILITY:
Inclusion Criteria:

* Patient who has provided written and informed consent
* Adult patient
* Patient undergoing cardiac surgery which is:

  1. Scheduled
  2. With bypass surgery
  3. Of the following types: aortic valve surgery, mitral valve surgery, tricuspid valve surgery, atrial myxoma, coronary artery bypass surgery, aortic surgery, combined surgery

Exclusion Criteria:

* Person not affiliated to national health insurance
* Person under legal protection (curatorship, guardianship)
* Person under court order
* Pregnant or breastfeeding woman
* Adult unable to express consent
* Patient already included once in the study
* Patient requiring emergency surgery within 24 hours
* Patients with hypersensitivity to local anesthetics or opiates or to any of the excipients in the products used
* Patients on antidepressants, neuroleptics such as non-selective MAOIs (iproniazid), selective A MAOI (moclobemide), selective B MAOI (selegiline) gabapentin (Neurontin®)
* Patients with an unprotected atrioventricular conduction disorder
* Patients with a prolonged QTc (> 450 ms) on preoperative ECG
* Patient with severe liver failure (PT< 30%)
* Patient suffering from respiratory failure (Long-term oxygen therapy patient except OSA)
* Patient with uncontrolled epilepsy
* Patient with preoperative cognitive dysfunction (MMS <24)
* Patient with intracranial hypertension
* Patient with chronic kidney failure (dialysis, creatinine > 200 μmol L-1)
* Patient with porphyria
* Patients treated with linezolid (Zyvoxid®)
* Patients with severe arterial hypotension (systolic BP<90 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one postoperative complication | 30 days post-surgery
  Post-operative complications:
  * postoperative neurological dysfunction
  * acute renal failure
  * acute respiratory failure
  * cardiovascular complications
  * death

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France